CLINICAL TRIAL: NCT06146088
Title: To Evaluate the Lot-to-lot Consistency of Immunogenicity, Safety, and Immune Persistence of Three Consecutive Commercial Manufacturing Batches of Inactivated Enterovirus 71 Vaccine (Human Diploid Cell) in Children Aged 6-35 Months in a Randomized, Blinded Study
Brief Title: Lot-to-lot Consistency Study of Three Commercial Batches of Enterovirus 71 Vaccine
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Institute of Medical Biology, Chinese Academy of Medical Sciences (Other)
Collaborators: Centers for Disease Control and Prevention, China (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: EV71-401
Record Dates: First submitted 2023-11-17; First posted 2023-11-24 (Actual); Last update posted 2024-01-03 (Actual); Status verified 2024-01

CONDITIONS: Hand, Foot and Mouth Disease
Keywords: Enterovirus 71; Inactivated enterovirus 71 vaccine
MeSH Terms: conditions — Hand, Foot and Mouth Disease

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Batch 1 (6-35 months old, 2 doses) (Experimental): Inactivated Enterovirus 71 Vaccine (human diploid cell) in children aged 6-35 months old on Day 0 and Day 30 approved by the National Institute for Food and Drug Control
  Interventions: Biological: EV71 Vaccine
- Batch 2 (6-35 months old, 2 doses) (Experimental): Inactivated Enterovirus 71 Vaccine (human diploid cell) in children aged 6-35 months old on Day 0 and Day 30 approved by the National Institute for Food and Drug Control
  Interventions: Biological: EV71 Vaccine
- Batch 3 (6-35 months old, 2 doses) (Experimental): Inactivated Enterovirus 71 Vaccine (human diploid cell) in children aged 6-35 months old on Day 0 and Day 30 approved by the National Institute for Food and Drug Control
  Interventions: Biological: EV71 Vaccine

INTERVENTIONS:
Biological: EV71 Vaccine — Inactivated enterovirus 71 vaccine (human diploid cell) of 3.0EU/0.5mL on Day 0,30

SUMMARY:
This study is a randomized, blinded study to evaluate the lot-to-lot consistency of immunogenicity, safety, and immune persistence of three consecutive manufacturing lots of EV71 vaccine, in 1500 children aged 6-35 months. The primary immunogenicity endpoint is the anti-EV71 neutralizing antibody geometric mean titer (GMT) 30 days after the final dose. The secondary immunogenicity endpoints are the geometric mean fold increases and seroconversion rates of anti-EV71 neutralizing antibodies 30 days after the final dose. The immune persistence endpoints are the seropositive rates as well as GMT of anti-EV71 neutralizing antibodies 12 and 24 months after the final dose. The safety endpoints are the number of adverse events/reactions within 30 minutes after each dose, the number of solicited adverse events/reactions within 7 days after each dose, the number of unsolicited adverse events/reactions within 30 days after each dose, and the number of serious adverse events (SAE) from the first dose to 6 months post the final dose.

DETAILED DESCRIPTION:
This study is a randomized, blinded study to evaluate the lot-to-lot consistency of immunogenicity, safety, and immune persistence of three consecutive manufacturing lots of EV71 vaccine, in children aged 6-35 months. The study is conducted to enroll 1500 healthy participants, including 600 infants aged 6-11 months, 600 toddlers aged 12-23 months, and 300 children aged 24-35 months. Eligibility will be assessed through medical history and physical examination. Participants from each age group will be randomly assigned to three different batch groups in a ratio of 1:1:1, that is, 500 participants in total will be in each lot arm, respectively.

All participants will receive an injection of the EV71 vaccine in the anterolateral midthigh or deltoid muscle of the upper arm on Day 0 and Day 30, respectively. The duration of interventions for each participant is approximately 1 month, thus, the duration of the immune persistence study for each participant is approximately 25 months.

For immunogenicity and immune persistence assessment, neutralizing antibodies against EV71 of all participants will be assessed on the first day (Day 0) before administration, 30 days after the final dose, and 12 and 24 months after the final dose, respectively.

For safety assessment, observation of adverse events (AE) from Day 0 to Day 30 after each dose of vaccination will be evaluated by diary or contact cards. Simultaneously, the serious adverse event (SAE) between the first dose of the vaccine to 6 months after the final dose will be evaluated by diary or contact cards, active reports, investigators' phone calls, or on-site visits. Meanwhile, participants will be observed at clinical sites for at least 30 minutes.

ELIGIBILITY:
Inclusion Criteria:

* Age Requirement: Children aged 6 to 35 months at the time of enrollment.
* Provision of legal Identification: Volunteers and their legal guardians or appointed representatives must provide valid legal identification documents.
* Informed Consent: Legal guardians or appointed representatives of volunteers must have the capacity to understand the informed consent document and the research process, voluntarily participate, sign the informed consent form, and be able to comply with the study's requirements and complete relevant visits on time.
* Temperature Requirement: Axillary body temperature prior to vaccination is less than 37.3°C.

Exclusion Criteria:

[First Dose Exclusion Criterions] Subjects meeting any of the following exclusion criteria will not be eligible for enrollment

* Allergic History: Subjects have a previous history of allergies to any component of the vaccine (e.g., aluminum hydroxide, glycine), or previous or suspected allergy to any vaccine or other serious adverse reaction (e.g., anaphylactic shock, laryngeal edema, anaphylactic purpura, thrombocytopenic purpura, local anaphylactic necrosis reaction, dyspnea, angioedema, systemic rash and/or urticaria, etc.).
* Vaccination History: Subjects received any inactivated vaccine or subunit vaccine within 7 days prior to the first dose of the investigational vaccine or any live attenuated vaccine within 14 days prior to the first dose of the investigational vaccine.
* Neurological and Mental Health: Subjects with a history or family history of convulsion, epilepsy, encephalopathy, and psychosis.
* Health Conditions: Subjects with known severe congenital malformation or developmental disorder (e.g., Down syndrome, sickle cell anemia, congenital neurological disorders).
* Acute Illness: Subjects have experienced acute illness (e.g., fever) or acute onset of chronic illness within 3 days before the first dose of investigational vaccine, or use of antipyretic, analgesic, or antiallergic drugs within 3 days before the first dose of the investigational vaccine.
* Coagulation Abnormalities: Subjects with genetic bleeding tendency, coagulopathy, or a history of bleeding disorders.
* Organ Removal History: Subjects have a history of surgical removal of the spleen or other vital immune organs for any reason.
* Blood Conditions: Subjects with blood loss (≥400mL) or receipt of blood transfusion, immune globulin (other than hepatitis B immune globulin), or blood products within 3 months prior to the first dose of the investigational vaccine.
* Drug Administration: Subjects use any investigational or unregistered product (drug, biological product, or device) within 3 months prior to the first dose of the investigational vaccine, or planned use during the study, except the investigational vaccine.
* Immune Therapy: Subjects have a treatment with immunosuppressive agents within 6 months before the first dose of the investigational vaccine, such as long-term treatment with systemic glucocorticoids (e.g., prednisone or a similar agent for more than 2 consecutive weeks within 6 months), but topical use (e.g., ointments, eye drops, inhalers, or nasal sprays) would be allowed.
* Previous history of receipt of other EV71 vaccines.
* Previous history of hand-foot-mouth disease.
* Immune-related Disease: Subjects have been diagnosed with an infectious disease that may interfere with the conduct or completion of the study (e.g., tuberculosis, viral hepatitis, human immunodeficiency virus infection, etc.).
* Investigators' Discretion: The final exclusion criterion is the investigator's discretion to determine whether a subject is suitable for participation in the study.

[Contraindication of the second dose of vaccine] Subjects meeting any of the following exclusion criteria will not be eligible for the second dose of the investigational vaccine

* Meeting allergic conditions that are mentioned in the First Dose Exclusion Criteria after the first dose.
* Severe Adverse Reactions: Subjects experienced serious adverse reactions after receiving the previous vaccine dose.
* Other Exclusion Reasons as Determined by the Investigator: The investigator determines other reasons for exclusion.

Ages: 6 Months to 35 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 1500 (Estimated)
Dates: Start 2023-11-25 (Actual); Primary Completion 2024-03-31 (Estimated); Study Completion 2026-07-15 (Estimated)

PRIMARY OUTCOMES:
Immunogenicity index-geometric mean titer (GMT) of neutralizing antibody | Day 30 after the second vaccination
  Neutralizing antibody assay will be performed using the neutralization and Microneutralization test method

SECONDARY OUTCOMES:
Immunogenicity index-geometric mean fold increase (GMFI) of neutralizing antibody | Between baseline and Day 30 after the second vaccination
  Neutralizing antibody assay will be performed using the neutralization and Microneutralization test method
Immunogenicity index-seroconversion rates of neutralizing antibody | Between baseline and Day 30 after the second vaccination
  Neutralizing antibody assay will be performed using the neutralization and Microneutralization test method.
  Seroconversion will be defined as a change from seronegative (<1:8) to seropositive (≥1:8), or ≥4-fold increase from baseline
Immunogenicity index-seropositive rates of neutralizing antibody | Day 30, 12 months, and 24 months after the second vaccination
  Neutralizing antibody assay will be performed using the neutralization and Microneutralization test method. Seropositive will be defined as the positive results with ties≥1:8
Safety index-incidence of adverse reactions/events | 0-30 minutes after the first dose vaccination
  Incidence of adverse reactions/events after the first dose vaccination
Safety index-incidence of adverse reactions/events | 0-30 minutes after the second dose vaccination
  Incidence of adverse reactions/events after the second dose vaccination
Safety index-incidence of adverse reactions/events | Day 0 to Day 7 after the first dose vaccination
  Incidence of solicited adverse reactions/events after the first dose vaccination
Safety index-incidence of adverse reactions/events | Day 0 to Day 7 after the second dose vaccination
  Incidence of solicited adverse reactions/events after the second dose vaccination
Safety index-incidence of adverse reactions/events | Day 0 to Day 30 after the first dose vaccination
  Incidence of unsolicited adverse reactions/events after the first dose vaccination
Safety index-incidence of adverse reactions/events | Day 0 to Day 30 after the second dose vaccination
  Incidence of unsolicited adverse reactions/events after the second dose vaccination
Safety index-incidence of serious adverse reactions/events | From the first dose to 6 months post the last dose of vaccination completed
  Occurrence of serious adverse reactions/events after vaccination

CONTACTS AND LOCATIONS:
Locations (4):
- China (4):
  - Chencang Center for Disease Prevention and Control, Baoji, Shaan XI
  - Ningqiang Center for Disease Prevention and Control, Hanzhong, Shaan XI
  - Fuping Center for Disease Prevention and Control, Weinan, Shaan XI
  - Jingyang Center for Disease Prevention and Control, Xianyang, Shaan XI

IPD SHARING:
Plan to Share IPD: No